CLINICAL TRIAL: NCT01836913
Title: Value of PET-CT in Radiation Treatment Planning for Patients With Esophageal Cancer
Acronym: RESPECT
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Johannes A. Langendijk, M.D., Ph.D., University Medical Center Groningen
Other Study IDs: RESPECT
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Cancer
Keywords: PET/CT; Esophageal cancer; Radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiotherapy for esophageal cancer: Patients with histology proven esophageal cancer who are planned for high dose radiotherapy with or without chemotherapy with or without surgery.

SUMMARY:
The RESPECT study is intended to prospectively assess the impact of PET/CT on the delineation of target volumes and to estimate the proportion of recurrences that could possibly be prevented by the use of PET/CT-based target volume, instead of CT-based. Patients will recieve radiotherapy using CT-based planning, but a PET/CT-based treatment plan will also be made. CT-based and PET/CT-based target volumes will be compared after treatment has been completed. If a locoregional recurrence takes place, the localisation will be compared to the CT-based and PET/CT based clinical target volumes (CTVs). If the local recurrence is located outside the CT-CTV but inside the PET/CT-CTV, the recurrence could possibly have been prevented with PET/CT-based radiotherapy.

DETAILED DESCRIPTION:
This is a prospective cohort study testing the hypothesis that in a proportion of patients, locoregional recurrence, observed at 6, 12 or 18 months after treatment, can be prevented if PET/CT-based treatment planning was used instead of CT-based treatment planning alone.

Patients eligible for the study will undergo definitive radiotherapy with or without concomitant chemotherapy with planning-CT based target volumes, either or not followed by surgery.

A planning-PET/CT will be made for research purposes only, and will be blinded for the treating physicians. This planning-PET/CT will not be used for actual treatment planning.

In case of neoadjuvant chemoradiation the response on this therapy will be analysed at pathologic evaluation of the esophageal specimen.

Routine follow up will be carried out every 6 months, using CT. In case of no locoregional recurrence and/or metastases, patients will be followed up to 18 months for study evaluation.

In case of distant metastases, patients will be censored if locoregional recurrence is excluded. When indicated, palliative treatment will be given.

In case of (suspicion of) locoregional recurrence, PET/CT-based recurrence analysis should be carried out with comparison and co-registration of CT-based and PET/CT-based target volumes.

ELIGIBILITY:
Inclusion Criteria:- Histologically proven adenocarcinoma or squamous cell carcinoma of the esophagus or GEJ

* Locally curable disease without distant metastases (M1b is excluded) (TNM clinical classification UICC 7th edition)
* Planned for high dose radiotherapy with or without chemotherapy with or without surgery
* Age ≥ 18 years;
* WHO performance status 0-2
* informed consent must be given according to ICH/EU GCP, and national/local regulations

Exclusion Criteria:- previous or concurrent malignancies (except basal cell carcinoma of the skin or in situ carcinoma of the cervix or superficial bladder cancer (pTa)) in the past five years

* Previous treatment
* Evidence of serious active infections
* any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven esophageal carcinoma who are planned for curative high dose radiotherapy with or without chemotherapy, with or without surgery.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Preventable locoregional recurrence by the use of PET/CT-based treatment planning, instead of CT-based | 18 months
  Proportion of patients with a locoregional recurrence, observed at 6, 12 or 18 months after treatment, can the recurrence be considered as possibly preventable if PET/CT-based treatment planning was used instead of CT-based treatment planning alone (located outside the CT-based CTV, but inside the PET/CT-based CTV)

SECONDARY OUTCOMES:
Differences in GTV, CTV and PTV for CT-based and PET/CT-based treatment planning | 6 months
  Differences in GTV (gross target volume), CTV and PTV (planning target volume) for CT-based and PET/CT-based treatment planning
Differences in dose distribution to OAR for CT and PET/CT-based treatment plans | 6 months
  Dose distribution in critical organs, including lung (mean lung dose, V20), heart (V30) and esophagus and calculation of NTCP values (Normal Tissue Complication Probability) comparing 3D-CRT and IMRT with and without PET/CT-based treatment planning
Percentage of patients who develop distant metastases after treatment | 18 months
  Percentage of patients who develop distant metastases after treatment
Cost-effectivity analyses | 24 months
  The costs of radiotherapy planning and treatment (surgical and/or chemoradiation), complications and recurrence-related treatment or the prevention thereof.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes A Langendijk, PhD, MD, Principal Investigator — University Medical Center Groningen, Department of Radiation Oncology; John Th Plukker, PhD, MD, Principal Investigator — University Medical Center Groningen, Department of Surgical Oncology
Locations (3):
- Netherlands (3):
  - RISO, Deventer, Overijssel
  - Medisch spectrum twente, Enschede, Overijssel
  - University Medical Center Groningen, Groningen, Provincie Groningen

REFERENCES:
- [Background] Muijs CT, Beukema JC, Pruim J, Mul VE, Groen H, Plukker JT, Langendijk JA. A systematic review on the role of FDG-PET/CT in tumour delineation and radiotherapy planning in patients with esophageal cancer. Radiother Oncol. 2010 Nov;97(2):165-71. doi: 10.1016/j.radonc.2010.04.024. Epub 2010 Jun 10. PMID 20541273
- [Result] Muijs CT, Pruim J, Beukema JC, Berveling MJ, Plukker JT, Langendijk JA. Oesophageal tumour progression between the diagnostic (1)(8)F-FDG-PET and the (1)(8)F-FDG-PET for radiotherapy treatment planning. Radiother Oncol. 2013 Mar;106(3):283-7. doi: 10.1016/j.radonc.2012.10.015. Epub 2012 Nov 27. PMID 23199654